CLINICAL TRIAL: NCT07188298
Title: Risk Factors, and Clinical Outcomes of Neonatal Anemia in the NICU of a Tertiary Care Hospital
Brief Title: Risk Factors and Clinical Outcomes of Neonatal Anemia in NICU
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Harris Ali, Assistant Lecturer, Assiut University
Other Study IDs: neonatal anemia
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hemolytic Disease of Newborn; Anemia of Neonates; Sepsis
MeSH Terms: conditions — Erythroblastosis, Fetal; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Risk Factors, and Clinical Outcomes of Neonatal Anemia in the NICU of a Tertiary Care Hospital

DETAILED DESCRIPTION:
Neonatal anemia is one of the most common hematological problems encountered in neonatal intensive care units (NICUs), particularly among preterm and very low birth-weight (VLBW) infants. It is defined as a hemoglobin (Hb) or hematocrit (Hct) concentration below the normal range for gestational and postnatal age, often necessitating clinical intervention to ensure adequate tissue oxygenation and prevent long-term neurodevelopmental consequences Anemia: Hb <13 g/dL in term newborns; Hb <12 g/dL in preterm neonates within the first week of life, according to WHO criteria The pathophysiology is multifactorial, involving both physiological and pathological processes. In preterm neonates, the condition known as anemia of prematurity (AOP) is primarily characterized by reduced erythropoietin production, shortened red blood cell (RBC) lifespan, and rapid postnatal growth that increases iron demand Globally, over 80% of extremely preterm infants (<28 weeks of gestation) require at least one RBC transfusion during their hospitalization . In Egypt, recent tertiary-level NICU data suggest that the prevalence of neonatal anemia among admitted preterm infants exceeds 60%, with many requiring multiple transfusions in the first month of life Major contributing factors include iatrogenic blood loss from frequent phlebotomy, insufficient iron stores at birth due to shortened gestation, hemolysis (immune or non-immune), and acute blood loss from perinatal events

ELIGIBILITY:
Inclusion Criteria:

* All live-born neonates admitted to the NICU within the first 24 hours of life.
* Both term and preterm infants.

Exclusion Criteria:

* Major congenital malformations
* Chromosomal abnormalities or genetic syndromes
* Neonates with a previous blood transfusion before study enrollment

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: neonates
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Understanding the local prevalence, associated factors, and outcomes of neonatal anemia | 1 year
  To determine the prevalence of neonatal anemia among neonates admitted to a tertiary care neonatal intensive care unit (NICU
  * To identify maternal, perinatal, and neonatal risk factors associated with neonatal anemia
  * To assess short-term outcomes, including length of hospital stay, need for blood transfusion, morbidity, and mortality

CONTACTS AND LOCATIONS:
Overall Officials: safwat abdelaziz, Study Director — Assiut University; m hamdy ghazaly, Study Director — Assiut University